CLINICAL TRIAL: NCT00815113
Title: Screening for Gastric Cancer in High-risk Population
Acronym: Stomach
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Niv, Director Department of Gastroenterology, Rabin Medical Center
Other Study IDs: RMC080000CTIL
Record Dates: First submitted 2008-12-25; First posted 2008-12-29 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; screening; high-risk; relatives; gastroscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: First degree relative of gastric cancer patient
- 2: Consecutive gastro-esophageal reflux patients

SUMMARY:
Introduction: Gastric cancer is the world's second largest cause of cancer related deaths. In the Western world, as well as in Israel, this malignancy is less prevalent than colorectal cancer, but has higher morbidity and mortality. First degree relatives of patients with gastric cancer have a 1.5-fold to 3-fold increased risk of developing gastric cancer themselves. In relatives of gastric cancer patients who are also carriers of a CagA positive strain of Helicobacter pylori, the risk is 8-fold. Mucosal atrophy, hypochlorhydria, high lymphoid follicle density, pan gastritis, and interleukin 1 β polymorphism are frequent in family members of gastric cancer patients and are associated with increased risk of the disease.

Aims:

1. To characterize the high risk individual for gastric cancer development.
2. To establish a screening plan for early detection and prevention of gastric cancer in first degree relatives of gastric cancer patients.
3. To validate new procedures for assessing risk factors for development of gastric cancer: gastric acid output, gastric mucin output, serum levels of pepsinogen I, pepsinogen II, gastrin B12, Helicobacter pylori status [serology, histology, urease test, 13C-urea breath test (13C-UBT)].
4. To assess genetic changes in the gastric mucosa of the screenees in comparison with gastric cancer patients and controls.

Methods:

We will approach 50 gastric cancer patients treated in Rabin Medical Center, and ask for their consent to approach first degree relatives for participating in the study. For each gastric cancer patient 4 relatives will be asked to signed an informed consent and undergo the study procedures. For each participant a matched control for age, sex and background diseases, out of consecutive gastro esophageal reflux disease (GERD) patients undergoing gastroscopy, will be asked to join the study. Thus, we will screen 50 gastric cancer patients, 200 first degree relatives of gastric cancer patients, and 200 controls.

DETAILED DESCRIPTION:
High Risk Population

First degree relatives of patients with gastric cancer have a 1.5-fold to 3-fold increased risk of developing gastric cancer themselves (Brenner H et al, Cancer 2000;88:274-9). In relatives of gastric cancer patients who are also carriers of a CagA positive strain of H. pylori, the risk is 8-fold. Mucosal atrophy, hypochlorhydria, high lymphoid follicle density, pangastritis, and interleukin 1 β polymorphism are frequent in family members of gastric cancer patients and are associated with increased risk of the disease (El-Omar EM et al, Gastroenterology 2000;118:22-30, Sepulveda A et al, Am J Gastroenterol 2002;97:1365-70).

Helicobacter Pylori - Carcinogen Number I

Helicobacter pylori is the main known carcinogen. The positive correlation between H. pylori infection and development of gastric cancer is well established and proved in prospective, controlled, studies, in Japan (Uemura N et al, N Engl J Med 2001;345:784-9, Fukase K et al, JAMA 2008;372:392-7).

Genetic changes

Specific changes (mutation in oncogens, LOH of tumor suppressor genes, deletion or insertion), different for intestinal or diffuse type gastric cancer, were described. Most of these pre-malignant changes happened on a background of long lasting chronic inflammation, following the cascade of atrophy, intestinal metaplasia, and dysplasia. Genetic syndromes are rare and families clustering of gastric cancer are usually attributed to common H. pylori infection. A family syndrome of gastric cancer due to germ-line mutation in E-cadherin has been described, and gastric cancer may be part of Lynch syndrome (HNPCC). Mutations and polymorphism of IL-1b and TNFa have been described in first degree relatives of gastric cancer patients, and considered predictive factors for cancer.

Screening for Gastric Cancer

Screening for gastric cancer gained popularity in Japan, where the disease is highly prevalent. This approach is not cost-effective in the Western word, where gastric cancer incidence is low, but still cost-effective in high-risk population: Helicobacter pylori infected people, first degree relatives of gastric cancer patients, patients with autoimmune atrophic gastropathy and pernicious anemia, families with HNPCC and patients who underwent partial gastrectomy. Since treatment for gastric cancer is not very effective and 5-year-survival is low, it is recommended to screen this population with periodic gastroscopy and biopsies. The finding of high grade dysplasia or early gastric cancer will enable early intervention and cure. In addition H. pylori may be diagnosed in gastric biopsies (direct evaluation in H&E, Giemsa or Genta staining, culture, PCR or urease rapid test), mucin secretion pattern may be assessed by immunohistochemistry with PAb's, MAb's or lectins, JCV TAg may be demonstrated by IMH or PCR).

Mucins in the Healthy Stomach and Gastric Cancer

Normal gastric mucus expresses the mucins MUC1, MUC5AC and MUC6 (Carrato C et al, Gastroenterology 1994;107:160-72). The development of gastric carcinoma is associated with changes in mucin expression, namely a decrease in MUC5AC and MUC6 and aberrant de novo expression of other MUCs (Ho SB et al, Cancer Res 1995;55:2681-90). Helicobacter pylori infection induces a wide range of changes in the gastric mucus. There is a reversible alteration of mucus glycosylation, which affects the protective function of the gastric mucins (Ota H et al, Virchows Arch 1998;433:419-26).

Screening for the High-Risk Phenotype

In addition to gastroscopy and histology, which are the gold standards for screening and prevention of gastric cancer, several other approaches, some of them are non-invasive, were suggested. Acid hyposecretion can be measured directly or indirectly, mucin output can be measured in gastric secretion collected by a naso-gastric tube and mucin species identified by dot-blot for gastric mucins (MUC5AC, MUC6 and MUC1), H. pylori status can be defined with 13C-UBT, serology or stool antigen test, pepsinogen I, pepsinogen II, gastrin and B12 can be measured in the serum. The combination of the procedures mentioned above may contribute to an accurate characterization of the high-risk individual, suitable for invasive procedure such as gastroscopy with biopsies.

Aims

1. To characterize the high risk individual for gastric cancer development
2. To establish a screening plan for early detection and prevention of gastric cancer in first degree relatives of gastric cancer patients.
3. To validate new procedures for assessing risk factors for development of gastric cancer: gastric acid output, gastric mucin output, serum levels of pepsinogen I, pepsinogen II, gastrin B12, H. pylori status (serology, histology, urease test, 13C-UBT).
4. To assess genetic changes in the gastric mucosa of the screenees in comparison with gastric cancer patients and controls

Subjects

We will approach 50 gastric cancer patients treated in Rabin Medical Center, and ask for their consent to approach first degree relatives for participating in the study. For each gastric cancer patient 4 relatives will be asked to signed an informed consent and undergo the study procedures. For each participant a matched control for age, sex and background diseases, out of consecutive GERD patients undergoing gastroscopy, will be asked to join the study. Thus, we will screen 200 first degree relatives of gastric cancer patients, and 200 controls.

Inclusion Criteria

1. First relative, man or woman, of gastric cancer patients.
2. Signed informed consent.
3. Age 18-60.

Exclusion Criteria

1. Severe back ground disease.
2. State after gastric surgery.
3. COPD, CHF, CRF and any disease with respiratory disturbances.
4. Deviation of the nasal septum, lack of venous access at the dorsum of the hand or any other technical problem prevents gastric acid collection or base excess evaluation.

Study design

This is a prospective, controlled, 4 days study. All procedures followed are in accordance with the ethical standards of the committee on human experimentation of the Rabin Medical Center, and in accordance with the Declaration of Helsinki. In the screening meeting the participant or the control will be told about the aims and nature of the study, and will be comprehensively informed about all procedures, anticipated results and risks. After agreeing to participate they will sign the informed consent. A medical history, family history and symptomatic questionnaire will be filled, and the participant will be scheduled for gastroscopy. After a night fast gastroscopy will be performed, biopsies will be taken as needed for the different protocols (see below). Then gastric acid output, mucin output and alkaline tide studies will be performed. Blood will be drawn for "gastro panel" of BioHit, routine blood tests, B12, CEA, CA19-9, and CAG A serology. In another day, 13CUBT and IFOBT will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. First relative, man or woman, of gastric cancer patients.
2. Signed informed consent.
3. Age 18-60.

Exclusion Criteria:

1. Severe back ground disease.
2. State after gastric surgery.
3. COPD, CHF, CRF and any disease with respiratory disturbances.
4. Deviation of the nasal septum, lack of venous access at the dorsum of the hand or any other technical problem prevents gastric acid collection or base excess evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: First degree relatives of gastric cancer patients
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Characterization of the high-rik individual for gastric cancer - "Gastric Cancer Phenotype" | 2 years

SECONDARY OUTCOMES:
Establish a screen plan for high-risk population for gastric cancer | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Niv, MD, Principal Investigator — RMC
Locations (1):
- Department of Gastroenterology, Rabin Medical Center, Petah Tikva, Israel